CLINICAL TRIAL: NCT06023667
Title: Self-Management Assistance for Recommended Treatement (SMART) App Randomized Control Trial
Brief Title: SMART-IBD App Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMART-IBD
Record Dates: First submitted 2023-07-28; First posted 2023-09-05 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Diseases; IBD; Crohn Disease; Ulcerative Colitis
Keywords: IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study PI, statistician, co-investigators, and all personnel who are involved in endpoint assessments will be blinded. Only study coordinators will have access to the assignment of each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART-IBD (Experimental): The SMART-IBD app consists of educational content, medication reminders, and weekly app engagement challenges. App users will participate in weekly challenges that focus on topics such as adherence, sleep, and diary usage. Participants in this arm will complete one month of run-in diaries, one month of diaries during intervention, and one month of diaries post-intervention.
  Interventions: Behavioral: SMART-IBD
- Attention Control (No Intervention): Participants in this arm will not receive any intervention content. Participants in this arm will complete one month of run-in diaries, one month of diaries during intervention and one month of diaries post-intervention.

INTERVENTIONS:
Behavioral: SMART-IBD — Daily medication and diary completion reminders are provided to participants. Additional educational content regarding self-management skills will be provided.
  Arms: SMART-IBD

SUMMARY:
The objective of this trial is to test whether a smartphone app, SMART-IBD, is effective in improving medication adherence and self-management skills in adolescents with IBD. The investigators will conduct a randomized control trial to compare a sample of 20 youth (ages 13-17) with IBD using an app that has educational content and medication reminders to 20 youth in an attention control group. The length of the intervention will include one month of baseline adherence data collection, one month of intervention, and one month of post-treatment adherence data collection.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with Crohn's disease, ulcerative colitis, or indeterminate colitis (collectively IBD)
* Prescribed at least one medication used to treat IBD, regardless of route of administration
* Access to internet or wi-fi or data plan and access to smartphone
* English fluency for patient and clinician

Exclusion Criteria:

* Diagnosis of pervasive developmental disorder in patient or caregiver as determined by medical chart review
* Diagnosis of serious mental illness (e.g., schizophrenia) in patient or caregiver as determined by medical chart review

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 3 months
  Medication adherence will be measured using electronic monitoring of medications indicated being taken in the SMART-IBD app

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States